CLINICAL TRIAL: NCT00887380
Title: A Randomised Comparison of Anastrozole Commenced Before and Continued During Adjuvant Radiotherapy for Breast Cancer Versus Anastrozole and Subsequent Anti-oestrogen Therapy Delayed Until After Radiotherapy.
Brief Title: STARS Breast Trial (Study of Anastrozole and Radiotherapy Sequencing)
Acronym: STARS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROG 08.06; ACTRN12610000307000 (Registry Identifier: ANZCTR)
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Timing of Radiotherapy; Local control
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Concurrent (Active Comparator): Investigational treatment: Anastrozole commenced before (Pre-radiotherapy commencement of anastrozole) and continued during radiotherapy.
  Interventions: Drug: Pre-radiotherapy commencement of anastrozole; Radiation: Radiotherapy
- Arm B: Sequential (Active Comparator): Standard Treatment: Anastrozole and subsequent anti-oestrogen therapy delayed until after radiotherapy (Post radiotherapy commencement of anastrozole)
  Interventions: Radiation: Radiotherapy; Drug: Post radiotherapy commencement of anastrozole

INTERVENTIONS:
Drug: Pre-radiotherapy commencement of anastrozole — Anastrozole: 1mg per day will be prescribed for 12 weeks. Commencing within 1 week of randomisation, to be administered from a min of 1 week before and a max of 4 weeks before commencement of radiotherapy and continued throughout radiotherapy. After 12 weeks administration of anastrozole according to trial regimen, anastrozole can be continued at the treating clinician's discretion and in accordance with the preference selected at the time of randomisation and stratification. The alternative options to long-term anastrozole are tamoxifen or cessation of anti-oestrogen therapy.
  Other Names: Arimidex
  Arms: Arm A: Concurrent
Radiation: Radiotherapy — Radiotherapy must commence within 1 month of randomisation. Radiotherapy planning and treatment is as per the protocol.
  Other Names: RT, Radiation Therapy
Drug: Post radiotherapy commencement of anastrozole — Anastrozole 1mg per day will be prescribed for 12 weeks after radiotherapy is completed. Anastrozole should commence within 1 week of the last fraction of radiotherapy and be continued for a total of 12 weeks. After 12 weeks administration according to the trial regimen, any subsequent hormone therapy is as for the concurrent arm.
  Other Names: Arimidex
  Arms: Arm B: Sequential

SUMMARY:
The purpose of this study is to determine whether starting anastrozole prior to radiotherapy, so that it is taken during radiotherapy, decreases local recurrence of breast cancer in post-menopausal women in comparison to waiting until after radiotherapy to commence anastrozole.

DETAILED DESCRIPTION:
Adjuvant radiotherapy is well established as the primary modality to enhance local control in breast cancer. The use of adjuvant hormone therapy such as tamoxifen has shown to improve local control to a relatively minor amount on its own and does enhance local control of adjuvant radiotherapy. There is, however, conflicting invitro and clinical data regarding the effects or different sequences on tamoxifen and radiotherapy in terms of both local control and enhancement of radiotherapy toxicities.

Aromatase inhibitors such as anastrozole are establishing themselves as a class of drug superior to tamoxifen for the control of estrogen dependent breast cancers and overall are better tolerated with the exception of greater bone loss.

As the key question is whether the sequencing of the aromatase inhibitor anastrozole alters local control by acting as an enhancer of the radiation breast cancer cell kill, it is therefore the aim of this study to compare 3 months of anastrozole prior to radiotherapy versus 3 months of anastrozole after radiotherapy with a specific objective of reducing the baseline ratio of in-field radiotherapy failure from 6% to 3%.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older
* Post total mastectomy or lumpectomy. All planned cancer resection surgery complete.
* Histologic or pathologic reports must verify either:

  * No tumour contacting the inked margin of surgically removed tissue, or
  * Focal involvement (<2mm front) if the margin is at the deep (posterior part) of the breast and the surgeon confirms that surgery extended to the deep fascia, or
  * Focal involvement (<2mm front) if the margin is superficial (anterior part of the breast or subcutaneous) and the surgeon confirms that surgery extended to the subcutis NB: In the case of focally involved deep or superficial margins, the medical records or multidisciplinary meeting notes or correspondence from the surgeon must indicate that the surgeon confirms the surgery extended to the deep fascia or subcutis as appropriate. Patients should routinely receive a lumpectomy bed boost in the conserved breast setting if there is focal superficial or focal deep involvement as defined above.
* Tumour oestrogen receptor and/or progesterone receptor positive (≥10% cells positive).
* Radiotherapy not yet commenced
* Planned radiotherapy dose prescribed to ICRU reference points in the irradiated breast / chest wall volumes at least the biological equivalent of 45 Gy in 25 fractions or more. (BED Gy4 ≥ 65, BED Gyx=D(1+n/x) where D=total dose, n=dose per fraction, x=alpha beta ratio, Gy4 selected as appropriate alpha-beta ratio for human breast cancer lines)
* An ECOG performance status score of 2 or less.
* Female and post menopausal shown by satisfying at least one of the following criteria (as per the ATAC study criteria16):

  * bilateral oophorectomy
  * age greater than 60
  * age 45-59 years with intact uterus and amenorrhoeic at least 12 months
  * Amenorrhoeic less than 12 months with follicle stimulating hormone (FSH) levels within the post menopausal range (including patients with amenorrhoea due to chemotherapy, LHRH use or who have had hormone replacement following hysterectomy) Note: it is recommended for women under the age of 45 who have been rendered menopausal by chemotherapy that they be enrolled onto the strata which switches to Tamoxifen after the initial 3 months of anastrozole.
* Is not receiving chemotherapy, or is receiving chemotherapy but the course will be completed at least 3 weeks prior to commencing radiotherapy
* Unilateral treatment
* Has provided written informed consent for participation in this trial

Exclusion Criteria:

* Previous radiotherapy to the area to be treated
* Previous invasive malignancy within 5 years of current breast cancer diagnosis with the exception of cervix in-situ or skin cancer other than melanoma.
* Patients with clinical evidence of metastatic disease.
* Previous hormonal breast cancer therapy.
* Ongoing hormone replacement therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2023 (Actual)
Dates: Start 2009-09-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To determine if commencement of anastrozole prior to radiotherapy results in improved local control compared to anastrozole commenced after radiotherapy. | 10 years post radiotherapy

SECONDARY OUTCOMES:
Rates of distant failure | 10 years post radiotherapy
Overall Survival | 10 years post radiotherapy
Normal tissue complications | 10 years post radiotherapy
Cosmesis | 10 years post radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Peter Graham, MBBS, Study Chair — Trans Tasman Radiation Oncology Group
Locations (34):
- Australia (31):
  - The Canberra Hospital, Canberra, Australian Capital Territory
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Genesis Cancer Care Hurstville, Hurstville, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Central West Cancer Service, Orange, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Riverina Cancer Centre, Wagga Wagga, New South Wales
  - Illawarra Cancer Care Centre, Wollongong, New South Wales
  - Alan Walker Cancer Centre, Darwin, Northern Territory
  - Genesis Cancer Care, Auchenflower, Queensland
  - Cairns ROQ, Cairns, Queensland
  - Genesis Cancer Care, Chermside, Queensland
  - The Townsville Hospital, Douglas, Queensland
  - Radiation Oncology Gold Coast, Gold Coast, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Radiation Oncology - Mater Centre, South Brisbane, Queensland
  - Genesis Southport, Southport, Queensland
  - St Andrew's Toowoomba Hospital, Toowoomba, Queensland
  - Genesis Care, Tugun, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Geelong Hospital, Geelong, Victoria
  - Genesis Cancer Care, Bunbury, Western Australia
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - Perth Radiation Oncology, Wembley, Western Australia
- New Zealand (3):
  - Auckland Hospital, Auckland
  - Christchurch Hopsital Oncology Sevice, Christchurch
  - Palmerston North, Palmerston North

REFERENCES:
- [Derived] Browne LH, Graham PH. Good intentions and ICH-GCP: Trial conduct training needs to go beyond the ICH-GCP document and include the intention-to-treat principle. Clin Trials. 2014 Dec;11(6):629-34. doi: 10.1177/1740774514542620. Epub 2014 Jul 14. PMID 25023199
- See also: Link to the TROG website where trial information can be found. — http://www.trog.com.au